CLINICAL TRIAL: NCT01192542
Title: Dispensing Evaluation of a New Galyfilcon A Prototype and Avaira Lenses
Brief Title: Pilot Evaluation of a New Galyfilcon A Lens Prototype and Enfilcon A Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CR-1636BE
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Results first posted 2014-01-17 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2016-05

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- galyfilcon A prototype lens/enfilcon A lens (Other): galyfilcon A prototype contact lens worn daily for 6-8 days first then enfilcon A contact lens worn daily for 6-8 days second.
  Interventions: Device: galyfilcon A prototype lens; Device: enfilcon A lens
- enfilcon A lens/galyfilcon A prototype lens (Other): enfilcon A contact lens worn daily for 6-8 days first then galyfilcon A prototype contact lens worn daily for 6-8 days second.
  Interventions: Device: galyfilcon A prototype lens; Device: enfilcon A lens

INTERVENTIONS:
Device: galyfilcon A prototype lens — Prototype silicone hydrogel contact lens
Device: enfilcon A lens — Marketed silicone hydrogel contact lens
  Other Names: Avaira® contact lens

SUMMARY:
The purpose of this study is to compare the visual acuity, limbal and bulbar redness of the new galyfilcon A prototype lenses against Avaira® lenses when worn as daily wear for seven (7) days.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a current spherical soft contact lens wearer and willing to wear the study lenses on a daily wear basis for the duration of the study.
* The subject's optimal vertexed spherical equivalent distance correction must be between -1.00 and - 5.00D.
* Any cylinder power must be ≤ -0.75D.
* The subject must have visual acuity best correctable to 20/25+3 or better for each eye.
* The subject must read and sign the Statement of Informed Consent.
* The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.

Exclusion Criteria:

* Ocular or systemic allergies or disease which might interfere with contact lens wear.
* Systemic disease or use of medication which might interfere with contact lens wear.
* Clinically significant (grade 3 or 4) corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear.
* Clinically significant (grade 3 or 4) tarsal abnormalities or bulbar injection which might interfere with contact lens wear.
* Any ocular infection.
* Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
* Pregnancy or lactation.
* Diabetes.
* Infectious diseases (e.g. hepatitis, tuberculosis) or an immuno-suppressive disease (e.g. HIV).
* Habitual contact lens type is toric, multifocal, or is worn as extended wear.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2010-08; Primary Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Pismo Beach, California
  - Warwick, Rhode Island
  - Fincastle, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 39 enrolled, with one screen failure prior to randomization, leaving 38 starting and completing the study.
Groups:
- Galyfilcon A Prototype Lens/Enfilcon A Lens: The galyfilcon A prototype contact lens worn daily for 6-8 days first then the enfilcon A contact lens worn daily for 6-8 days second.
- Enfilcon A Lens/Galyfilcon A Prototype Lens: The enfilcon A contact lens worn daily for 6-8 days first then the galyfilcon A prototype contact lens worn daily for 6-8 days second.
Period: Period 1
Arm/Group | Galyfilcon A Prototype Lens/Enfilcon A Lens | Enfilcon A Lens/Galyfilcon A Prototype Lens
Started | 18 | 20
Completed | 18 | 20
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Galyfilcon A Prototype Lens/Enfilcon A Lens | Enfilcon A Lens/Galyfilcon A Prototype Lens
Started | 18 | 20
Completed | 18 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline summary was conducted on all enrolled subjects.
Groups:
- All Subjects: All subjects who enrolled in the study.
Arm/Group | All Subjects
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (6.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Monocular Visual Acuity Assessment
Description: Snellen monocular visual acutity (VA) assessed by the Investigator and was converted to the LogMAR scale.
Time Frame: Post lens insertion (baseline)
Population: Analysis was conducted on subjects who were enrolled, randomized, and successfully completed the study.
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: eyes
Groups:
- Galyfilcon A Prototype Lens: Prototype silicone hydrogel lens.
- Enfilcon A Lens: Marketed silicone hydrogel lens.
Arm/Group | Galyfilcon A Prototype Lens | Enfilcon A Lens
Number analyzed (Participants) | 38 | 38
Number analyzed (eyes) | 76 | 76
logMAR | -0.05 (0.0317) | -0.04 (0.0317)
Statistical Analysis 1: Comparison: Galyfilcon A Prototype Lens vs Enfilcon A Lens; The alternative hypothesis is the monocular visual acuity of the galyfilcon A prototype lens is non-inferior to that of the enfilcon A lens; Test type: Non-Inferiority or Equivalence — The non-inferiority margin of 0.05 (1/2 LogMAR line) was used; Mixed Models Analysis; Comparisons between two lenses were carried out using 95% confidence intervals (CI) constructed for least-square mean differences; Least-square mean difference = -0.009, 95% CI 2-sided [-0.022 to 0.003], Standard Error of Mean 0.0064 — The mean difference is calculated as: Test lens - Control lens

2. Secondary Outcome: Limbal Redness of Grade 3 or Above
Description: Limbal redness was assessed using a 5-point slit lamp classification scale (5-Worst, 0-None). Only those eyes with limbal redness grade >= 3 were reported for purposes of this analysis. Grades 3 -5 are considered to be part of the adverse events reporting.
Time Frame: After 6-8 days of lens wear
Population: Analysis was conducted on subjects who successfully completed the study.
Measure: Number; unit: Subject Eyes
Units Other Than Participants: Eyes
Groups:
- Galyfilcon A Prototype Lens: Prototype silicon hydrogel contact lens.
Arm/Group | Galyfilcon A Prototype Lens | Enfilcon A Lens
Number analyzed (Participants) | 38 | 38
Number analyzed (Eyes) | 76 | 76
Subject Eyes | 0 | 0

3. Secondary Outcome: Bulbar Redness of Grade 3 or Above
Description: Bulbar redness was assessed using a 5-point slit lamp classification scale (5-Worst, 0-None). Only those eyes with bulbar redness grade >= 3 were reported for purposes of this analysis. Grades 3 -5 are considered to be part of the adverse events reporting.
Time Frame: After 6-8 days of lens wear
Population: Analysis was conducted on subjects who successfully completed the study.
Measure: Number; unit: Subject Eyes
Units Other Than Participants: Eyes
Arm/Group | Galyfilcon A Prototype Lens | Enfilcon A Lens
Number analyzed (Participants) | 38 | 38
Number analyzed (Eyes) | 76 | 76
Subject Eyes | 0 | 0

4. Primary Outcome: Binocular Visual Acuity
Description: Snellen binocular visual acuity assessed by the Investigator and was converted to the LogMAR scale. A value <0 implies clinically positive results, a value >0 implies clinically negative results
Time Frame: Post lens insertion (baseline)
Population: Analysis was conducted on subjects who enrolled, were randomized, and successfully complete the study per protocol.
Measure: Least Squares Mean (Standard Error); unit: LogMAR
Arm/Group | Galyfilcon A Prototype Lens | Enfilcon A Lens
Number analyzed (Participants) | 38 | 38
LogMAR | -0.08 (0.032) | -0.08 (0.032)
Statistical Analysis 1: Comparison: Galyfilcon A Prototype Lens vs Enfilcon A Lens; The alternative hypothesis is the binocular visual acuity of the galyfilcon A prototype lens is non-inferior to that of the enfilcon A lens; Test type: Non-Inferiority or Equivalence — The non-inferiority margin of 0.05 (1/2 LogMAR line) was used; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Least-square mean difference = 0, 95% CI 2-sided [-0.018 to 0.018], Standard Error of Mean 0.0091

ADVERSE EVENTS:
Time Frame: Adverse events were recorded when the subjects were exposed to the Investigational lenses.
Groups:
- All Subjects: All subjects who exposed to the Investigation lenses.
Arm/Group | All Subjects
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No